CLINICAL TRIAL: NCT07279324
Title: Pilot Study on the Safety and Efficacy of Kelulut Honey Eyedrops for Dry Eye Disease
Brief Title: Safety and Efficacy of Kelulut Honey Eyedrops in Dry Eye Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Shahidatul Adha Mohamad, Dr., Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USM-KHED-2025-01
Record Dates: First submitted 2025-11-30; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Dry Eye Disease (DED); Dry Eye Syndrome (DES); Dry Eye Symptoms
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: A randomized, parallel, three-arm pilot study comparing the safety and preliminary efficacy of Kelulut honey eyedrops at three concentrations (12.5%, 25%, and 50%) over a 1-month treatment period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is masked to participants, care providers, investigators, and outcome assessors. The Kelulut honey eyedrops will be dispensed in identical sterile droppers labeled only with coded allocation numbers. The pharmacist preparing and dispensing the formulations is the sole unmasked individual. Investigators and assessors will remain blinded throughout the intervention period and until all data collection is complete. Unmasking will occur only after database lock, when the pharmacist releases the allocation code for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- KHED 12.5% (Experimental): Participants in this arm will use Kelulut honey eyedrops formulated with Kelulut honey derived from stingless bees (Trigona spp.) at a concentration of 12.5%. The eyedrops will be administered three times daily for 1 month, in addition to the participant's usual dry eye treatments. Safety, tolerability, and changes in tear film parameters will be assessed.
  Interventions: Drug: Kelulut Honey Eyedrop 12.5%
- KHED 25% (Experimental): Participants in this arm will use Kelulut honey eyedrops formulated with Kelulut honey derived from stingless bees (Trigona spp.) at a concentration of 25%. The eyedrops will be administered three times daily for 1 month, in addition to the participant's usual dry eye treatments. Safety, tolerability, and changes in tear film parameters will be assessed.
  Interventions: Drug: Kelulut Honey Eyedrop 25%
- KHED 50% (Experimental): Participants in this arm will use Kelulut honey eyedrops formulated with Kelulut honey derived from stingless bees (Trigona spp.) at a concentration of 50%. The eyedrops will be administered three times daily for 1 month, in addition to the participant's usual dry eye treatments. Safety, tolerability, and changes in tear film parameters will be assessed.
  Interventions: Drug: Kelulut Honey Eyedrop 50%

INTERVENTIONS:
Drug: Kelulut Honey Eyedrop 12.5% — KHED 12.5% is sterile ophthalmic solution containing Kelulut honey derived from stingless bees (Trigona spp.) at a concentration of 12.5%. Participants will instill one drop in each eye three times daily for 30 days, in addition to their usual dry eye treatments.
  Arms: KHED 12.5%
Drug: Kelulut Honey Eyedrop 25% — KHED 25% is sterile ophthalmic solution containing Kelulut honey derived from stingless bees (Trigona spp.) at a concentration of 25%. Participants will instill one drop in each affected eye three times daily for 30 days, in addition to their usual dry eye treatments.
  Arms: KHED 25%
Drug: Kelulut Honey Eyedrop 50% — KHED 50% is sterile ophthalmic solution containing Kelulut honey derived from stingless bees (Trigona spp.) at a concentration of 25%. Participants will instill one drop in each affected eye three times daily for 30 days, in addition to their usual dry eye treatments
  Arms: KHED 50%

SUMMARY:
The goal of this clinical trial is to learn whether Kelulut honey eyedrops are safe and helpful in treating dry eye disease in adults. It will also learn about any side effects that may occur with the use of Kelulut honey eyedrops.

This Kelulut honey eyedrops are sterile ophthalmic solutions formulated with honey derived from stingless bees (Trigona spp.) at concentrations of 12.5% 25% and 50%. The eyedrop formulations are prepared according to a standardized laboratory protocol to ensure sterility, stability, and suitability for ocular use. Full formulation details are proprietary but can be provided to the ethics committee or regulatory authorities upon request.

The main questions this clinical trial aims to answer are:

1. Does Kelulut honey improve tear film stability and dry eye symptoms?
2. Are Kelulut honey eyedrops safe and well tolerated on the ocular surface?

Researchers will compare different concentrations of Kelulut honey eyedrops to determine which concentration provides the best balance of safety and clinical benefit.

Participants will:

1. Use Kelulut honey eyedrops (12.5%, 25%, or 50%) three times daily for 1 month, in addition to continuing their usual dry eye treatments.
2. Attend scheduled follow-up visits (on week 2 and week 4) for eye examinations and dry eye assessments (e.g., TBUT, ocular surface staining, Schirmer test, and OSDI).
3. Report any changes in symptoms or any discomfort, including stinging, redness, irritation, or other adverse effects experienced during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50 years at the time of consent.
2. Clinical diagnosis of dry eye disease in at least one eye, based on symptoms and clinical signs (Symptomatic dry eye, defined as an OSDI score ≥ 13; objective evidence of tear film instability, such as TBUT < 10 seconds in at least one eye)
3. Participants may be Treatment-naïve, OR on stable dry eye treatment for at least 2 weeks before enrollment.
4. Willing to use Kelulut honey eyedrops three times daily for 1 month as instructed.
5. Able and willing to attend all study visits (Baseline, Week 2, Week 4).

Exclusion Criteria:

1. Known allergy or hypersensitivity to honey, bee products, or any component of the study formulations.
2. Active ocular infection or inflammation (e.g., infectious conjunctivitis, keratitis, uveitis).
3. Severe allergic conjunctivitis or other ocular surface diseases
4. Significant meibomian gland dysfunction or blepharitis
5. Ocular surgery or laser procedures within the past 6 months.
6. Use of topical ocular medications other than lubricants within the past 30 days
7. Contact lens wear within 1 week prior to baseline or expected during the study.
8. Punctal plugs or other lacrimal procedures within the last 3 months.
9. Systemic diseases that significantly affect the ocular surface and are unstable or uncontrolled (e.g., uncontrolled Sjögren's, uncontrolled rheumatoid arthritis, uncontrolled diabetes).
10. Participation in another clinical trial or receipt of an investigational product within the past 30 days.
11. Pregnant or breastfeeding women, or those planning pregnancy during the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in Corneal Fluorescein Staining Score | Baseline, Week 2 and Week 4
  Corneal staining will be assessed using slit lamp biomicroscopy and graded using the National Eye Institute (NEI) scale. The cornea is divided into five zones (central, superior, inferior, nasal, temporal), each scored from 0 to 3 based on dot count:
  0 = no staining
  1. = 1-5 punctate dots
  2. = 6-30 punctate dots
  3. = >30 dots or coalescent staining

SECONDARY OUTCOMES:
Changes in Tear Break-Up Time (TBUT) | Baseline, Week 2 and Week 4.
  TBUT will be measured after fluorescein instillation. The interval between the last blink and the first appearance of a dry spot on the cornea will be recorded. Three readings will be averaged. Longer TBUT indicates better tear film stability.
Changes in Ocular Surface Disease Index (OSDI) score | Baseline, Week 2 and Week 4.
  The OSDI is a short 12-question survey that asks how often you experience dry eye symptoms and how much they affect your daily activities. Each question is scored from 0 ("none of the time") to 4 ("all of the time"). The total score ranges from 0 to 100, with higher scores meaning more severe dry eye symptoms.
Schirmer I Test Value | Baseline, Week 2 and Week 4
  Schirmer I test will be performed to measure aqueous tear production. A sterile strip will be placed in the lower eyelid, and the length of strip wetting in millimeters will be recorded after 5 minutes.

OTHER OUTCOMES:
Conjunctival Hyperaemia Score | Baseline, Week 2 and Week 4.
  Bulbar conjunctival hyperemia will be graded using a 0-3 scale (0 = none, 3 = severe).
Subjective Ratings of Comfort | Baseline, Week 2 and Week 4.
  Participants will rate their eye comfort using a standardized scale from 0 to 10, where 0 means "unacceptable/very poor comfort" and 10 means "excellent comfort."

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Pakar Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No